CLINICAL TRIAL: NCT01461668
Title: Retapamulin for Reducing MRSA Nasal Carriage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Huang, Director of Epidemiology and Infection Prevention, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OCRT10049
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
Keywords: MRSA; MRSA resistant to mupirocin
MeSH Terms: interventions — retapamulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retapamulin (Experimental): Participants in this arm will be instructed to complete a decolonization regimen that will involve a 5-day application of retapamulin with follow up bilateral nares swab one week following completion of therapy (~D12) to assess clearance. If follow up swabs are positive for MRSA, patients will be given a second course of the same agent (retapamulin) to begin one week following swab collection (~D19-23) so that up to two decolonization attempts will be made. A final set of bilateral nares swabs will be obtained from all subjects six weeks from the completion of initial treatment (~D47).
  Interventions: Drug: Retapamulin
- Placebo (Placebo Comparator): Participants in this arm will be instructed to complete a decolonization regimen that will involve a 5-day application of a placebo with follow up bilateral nares swab one week following completion of therapy (~D12) to assess clearance. If follow up swabs are positive for MRSA, patients will be given a second course of the same agent (placebo) to begin one week following swab collection (~D19-23) so that up to two decolonization attempts will be made. A final set of bilateral nares swabs will be obtained from all subjects six weeks from the completion of initial treatment (~D47).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retapamulin — Two times a day for 5 days
  Other Names: Altabax
  Arms: Retapamulin
Drug: Placebo — Two times a day for 5 days
  Arms: Placebo

SUMMARY:
The investigators will conduct a randomized placebo-controlled double-blinded study of nasal decolonization with retapamulin vs. placebo for the eradication of MRSA nasal carriage among adult carriers with low-level (MIC 8-256) and high-level mupirocin resistant (MIC >256) strains.

Objectives:

1. To determine the percent of intervention vs. control patients with successful MRSA nasal decolonization as determined by bilateral nares swabs following a 5-day twice-a-day regimen of retapamulin.
2. To determine the time to decolonization based upon interim and final bilateral nares swabs.
3. To determine the acceptability of retapamulin by surveying participants about their experience and adverse events experienced during this study.

The duration of participant follow-up is expected to last up to 7 weeks.

This study will evaluate the safety and effectiveness of Altabax (retapamulin) during decolonization of MRSA carriers with mupirocin-resistant strains, stratified by low-level and high-level resistance to mupirocin. Mupirocin resistance is increasingly common and there is no approved substitute topical agent for decolonization of the MRSA nasal reservoir.

DETAILED DESCRIPTION:
This study will evaluate the utility of retapamulin, a topical ointment FDA approved for skin infection, as a novel agent for MRSA decolonization and prevention of healthcare-associated MRSA infection. Retapamulin is a first-in-class semi-synthetic pleuromutilin antibiotic that inhibits protein synthesis by interacting with the bacterial ribosome 50S subunit. It received FDA approval in 2007 for the topical treatment of impetigo in adults and pediatric patients.

We propose to evaluate retapamulin as an investigational agent for the nasal decolonization of MRSA carriers whose strains demonstrate low-level and high-level resistance to mupirocin. Mupirocin resistance is increasingly common and there is no approved substitute topical agent for decolonization of the MRSA nasal reservoir.

We will conduct a randomized placebo-controlled double-blinded study of nasal decolonization with retapamulin vs. placebo for the eradication of MRSA nasal carriage among adult carriers with low-level (MIC 8-256) and high-level mupirocin resistant (MIC >256) strains. Randomization will be stratified by low vs high level resistance.

Consenting adult (at least 18 years old) subjects will be randomized to 1% retapamulin or placebo ointment intra-nasally twice a day for 5 days (D1-5) with follow up bilateral nares swab one week following completion of therapy (~D12) to assess clearance. If follow up swabs are positive for MRSA, patients will be given a second course of the same agent (retapamulin or placebo) to begin one week following swab collection (~D19-23) so that up to two decolonization attempts will be made. A final set of bilateral nares swabs will be obtained from all subjects six weeks from the completion of initial treatment (~D47).

Consenting adult (at least 18 years old)subjects will be given retapamulin or placebo. At the time of recruitment, all subjects will complete a detailed survey administered by trained research staff. This survey will include questions related to self care, home hygiene practices, and known risk factors for MRSA acquisition. Subject follow up will include repeat bilateral nares swabs and follow up surveys related to compliance, experience (side effects/concerns) with the assigned regimen, and ongoing risk factors will occur either during a home visit (or facility visit if the patient is admitted to a hospital or nursing home at the time of the required visit) or at the University of California Irvine (UCI) Institute for Clinical and Translational Science (ICTS), a Clinical and Translational Science Award (CTSA) site which provides clinic visit support for pilot studies.

Outcomes will include successful nares decolonization at the end of the follow up period (D47). We will detail the sequence of clearance or re-colonization based upon the two follow up nares swabs, as well as any adverse events, which are expected to be related to local irritation in a small percent of subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have a type of MRSA that is resistant to mupirocin (a drug used to treat MRSA)

Exclusion Criteria:

* Allergic to retapamulin
* Unable to use retapamulin via your nose (i.e. nose surgery, etc.)
* Are pregnant and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Huang, MD, MPH, Principal Investigator — University of California, Irivne - School of Medicine
Locations (1):
- University of California, Irivne, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were identified from MRSA samples tested for Mup-R from the UC Irvine Medical Center microbiology lab and from samples from participants who completed a separate clinical trial. Of 294 patients found to have mupirocin resistant isolates, 53 were consented and randomized. Three dropped out prior to any intervention.
Period: Overall Study
Arm/Group | Retapamulin | Placebo
Started | 27 | 26
Completed | 25 | 25
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Number of participant totals reflect total subjects included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Retapamulin | Placebo | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (16.9) | 59.0 (16.2) | 59.7 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With MRSA Clearance
Description: Proportion of participants with MRSA clearance at the end of the follow up period
Time Frame: 47 days
Population: The total number of participants analyzed include those that completed the study (through day 47).
Measure: Count of Participants; unit: Participants
Arm/Group | Retapamulin | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 8 | 4
Statistical Analysis 1: Comparison: Retapamulin vs Placebo; Test type: Superiority; p = 0.320, Fisher Exact; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.08 to 1.86] — Confidence interval for the odds ratio is based upon the inversion Fisher's exact test

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Retapamulin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Recruitment challenges from low yield of mupirocin-resistant MRSA. Trial suspended when funding concluded. Extensive efforts to acquire new sites and new funding to extend trial requirement were unsuccessful. Trial was closed and analysis completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-01-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT01461668/Prot_000.pdf
  • Statistical Analysis Plan (2011-10-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT01461668/SAP_001.pdf